CLINICAL TRIAL: NCT01343433
Title: Influence of Bright Light Therapy on Delirium in Patients at the Intensive Care Unit: a Pilot-study
Brief Title: Influence of Light Therapy on Confusion in Patients at the Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: J.I. van der Spoel, Onze Lieve Vrouwe Gasthuis
Other Study IDs: D-3101-4
Record Dates: First submitted 2011-04-25; First posted 2011-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Delirium; Intensive Care Unit Syndrome
Keywords: Delirium; Intensive Care Unit Syndrome; Bright light therapy; Intensive Care Unit
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Chamber allocation will determine which patient receives bright light therapy. We selected four patient chambers at the Intensive Care Unit, each with the capacity of two patient beds. In two chambers patients will receive bright light therapy. Patients in the other two rooms are only exposed to environmental light
- Treatment group (bright light therapy): Chamber allocation will determine which patient receives bright light therapy. We selected four patient chambers at the Intensive Care Unit, each with the capacity of two patient beds. In two chambers patients will receive bright light therapy. During our study, light therapy will be applied with instrument 'Litepod' (manufactured by Goodlite, Donker Curtiusstraat 7/407, Amsterdam), which gives an intensity of 10000 lux at a distance of 22 centimetres.Patients will receive bright light therapy for three hours in the morning, from eight o'clock till eleven o'clock.

SUMMARY:
Our purpose of this study is to determine whether bright light therapy is effective for reducing the incidence and the duration of delirium compared to the usual treatment in patients at the Intensive Care Unit. Our hypothesis is that bright light therapy is effective for reducing the incidence and duration of delirium in patients at the Intensive Care Unit

Patients will be assigned to a chamber with or without bright light therapy. This assignment is based on occupation of ICU beds and availability of nurses and is therefore independent from patients characteristics. Patients will be included following the inclusion criterion and exclusion criteria. Patients assigned to a chamber with bright light therapy will receive light therapy for three hours in the morning, from eight o'clock till eleven o'clock. The Confusion Assessment Method-score (CAM-score) and the Richmond Agitation Sedation Scale-score (RASS-score) will be performed three times at one day by ICU nurses, this is according to the existing routine. Besides this, an extra CAM-score and a clinical assessment will be performed once a day by a trained non-clinician, to determine the presence of delirium. The use of sedatives, haldol and fixation will be registered to determine the occurrence, duration and severity of delirium. Eventually the most important outcomes will be the clinical assessment of the patients, the CAM-score and the use of haldol. The primary outcome of this study is the duration of delirium, defined in number of days.

DETAILED DESCRIPTION:
Intensive Care patients experience severe alterations of sleep. They may develop a circadian rhythm sleep disorder, characterized by an irregular sleep/wake pattern. The presence of abnormal sleep/wake cycles may be a risk factor for delirium, which would link it to higher morbidity, mortality and longer ICU stay. Bright light therapy is the treatment of choice for circadian rhythm sleep disorders and may be helpful in handling delirium. The objective of this study is to determine whether bright light therapy is effective for reducing the incidence and duration of delirium in the Intensive Care Unit.

This is a prospective, single center cohort investigation by witch the influence of bright light therapy on the incidence and duration of delirium will be examined and compared with environmental light. This study will take place at the ICU of the OLVG, a level three ICU with 24 beds in a teaching hospital.

Patients will be assigned to a chamber with or without bright light therapy. This assignment is based on occupation of ICU beds and availability of nurses and is therefore independent from patients characteristics. All patients of 18 years and older who will be admitted to the Intensive Care Unit of the Onze Lieve Vrouwe Gasthuis, Amsterdam can be included in the study. Patients diagnosed with bipolar disorder will be excluded from participation. Other exclusion criteria are the use of an antipsychotic drug in the home environment, temporary or permanent loss of total vision and participation in this study during a previous admission to the Intensive Care Unit.

Patients assigned to a chamber with bright light therapy will receive light therapy for three hours in the morning, from eight o'clock till eleven o'clock. The Confusion Assessment Method-score (CAM-score) and the Richmond Agitation Sedation Scale-score (RASS-score) will be performed three times at one day by ICU nurses, this is according to the existing routine. Besides this, an extra CAM-score and a clinical assessment will be performed once a day by a trained non-clinician, to determine the presence of delirium. The use of sedatives, haldol and fixation will be registered to determine the occurrence, duration and severity of delirium. Eventually the most important outcomes will be the clinical assessment of the patients, the CAM-score and the use of haldol.

At the Intensive Care Unit of the Onze Lieve Vrouwe Gasthuis, Amsterdam, light therapy is used by nurses for optimizing the light intensity in their work environment, for their own well being and for the prevention of sleep disturbances. The light therapy is also randomly used for the treatment of Intensive Care patients, though the effectiveness and functionality have not been a subject of investigation. Our purpose of this study is to determine whether bright light therapy is effective for reducing the incidence and the duration of delirium in the Intensive Care Unit. The primary outcome of this study is the duration of delirium, defined in number of days. This will be derived from the clinical assessments and the CAM-scores, performed by the trained non-clinician.

ELIGIBILITY:
Inclusion criterion:

* Age: a minimum age of 18 years

Exclusion criteria:

* Psychiatric comorbidity: bipolar disorder
* The use of an antipsychotic drug in the home environment
* Participation in this study during a previous admission to the ICU
* Temporary or permanent loss of total vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of 18 years and older who will be admitted to the Intensive Care Unit of the Onze Lieve Vrouwe Gasthuis, Amsterdam can be included in the study. This is a medical surgical level three ICU with 24 beds. There are over 90 specialised ICU nurses laborious in this ICU. An average of 1500 patients a year is admitted, of which 750 from the cardiothoracic surgical department.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Duration of delirium, defined in days | After 10 weeks
  The primary outcome of this study will be the duration of delirium, defined in number of days. This will be derived from the clinical assessments and CAM-scores, performed by the trained non-clinician.

SECONDARY OUTCOMES:
Incidence of delirium in the patient group receiving bright light therapy and in the group receiving environmental light | After 10 weeks
CAM-scores of the ICU nurses | After 10 weeks
  The Confusion Assessment Method-ICU is the most accurate diagnostic instrument to detect delirium in hospitalized patients and is the only instrument validated for detecting delirium in mechanically ventilated patients. These scores are already determined three times at one day by Intensive Care nurses.
Dosage of haloperidol use in delirious patients receiving bright light therapy and those receiving environmental light | After 10 weeks
  The dosage of haldol use will be registered to determine the presence and duration of delirium
Duration of haldol use in delirious patients receiving bright light therapy and those receiving environmental light | After 10 weeks
  The duration of haldol use will be registered to determine the presence and duration of delirium
Mortality of delirious patients in the ICU and in the hospital, comparing those who receive bright light therapy with those who receive environmental light | After 10 weeks
  We are interested in variables that could be influenced by the presence of delirium, including mortality.
Duration of mechanical ventilation in delirious patients receiving bright light therapy and those receiving environmental light | After 10 weeks
  We are interested in variables that could be influenced by the presence of delirium, including duration of mechanical ventilation
Duration of admission of delirious patients in the ICU and in the hospital, comparing those who receive bright light therapy with those who receive environmental light | After 10 weeks
  We are interested in variables that could be influenced by the presence of delirium, including the duration of admission
Duration of admission in the ICU and in the hospital, comparing those who receive bright light therapy with those who receive environmental light | After 10 weeks
  We are interested in variables that could be influenced by the presence of delirium, including the duration of admission

CONTACTS AND LOCATIONS:
Overall Officials: J.I van der Spoel, MD, Principal Investigator — Onze Lieve Vrouwe Gasthuis
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands